CLINICAL TRIAL: NCT04441320
Title: Efficacy and Safety of Coated Metal Ureteral Stent in the Treatment of Radiation Induced Ureteral Stricture, A Prospective, Mutlcenter and Controlled Study
Brief Title: Coated Metal Ureteral Stent in the Treatment of Radiation Induced Ureteral Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Huhao, Associate Professor, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO-02
Record Dates: First submitted 2020-06-14; First posted 2020-06-22 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Ureteral Stricture; Hydronephrosis; Radiation Exposure
Keywords: radiation induced ureteral stricture; coated metal ureteral stent; safety; efficacy
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMUS group (Experimental): Coated metal ureteral stent is indwelled.
  Interventions: Device: Coated metal ureteral stent(CMUS)
- DJS group (Other): Double-J stent is indwelled
  Interventions: Device: Double-J stent(DJS)

INTERVENTIONS:
Device: Coated metal ureteral stent(CMUS) — Coated metal ureteral stent aims to treat the patients with refractory ureteral stricture, such as radiation induced ureteral stricture. In this study, CMUS is indwelled to observe the efficacy and safety in the treatment of radiation induced ureteral stricture compared with Double-J stent.
  Arms: CMUS group
Device: Double-J stent(DJS) — Double-J stent is commonly used for treatment of kinds of ureteral stricture. In this study, DJS is indwelled as a controlled group.
  Arms: DJS group

SUMMARY:
A prospective, multicenter and controlled study to observe the efficacy and safety of coated metal ureteral stent in the treatment of radiation induced ureteral stricture.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ureteral stricture and hydronephrosis.
2. Previous history of radiation therapy.
3. Must be able to tolerate surgery.

Exclusion Criteria:

1. Combine with hypertonic neurogenic bladder (except for patients with long-term indwelling catheter).
2. Colon resection surgery patients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patency rate | Up to 36 months
  Number of patients evaluated with hydronephrosis
Indwelling time | Up to 36 months
  Number of months of the implant in the ureter
Device related serious adverse events | Up to 36 months
  Number of device related serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Peiking university people's hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No